CLINICAL TRIAL: NCT05223413
Title: REmote iSchemic condItioning in Lymphoma PatIents REceiving ANthraCyclinEs
Acronym: RESILIENCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RESILIENCE-H2020
Record Dates: First submitted 2021-12-20; First posted 2022-02-04 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-05

CONDITIONS: Anthracycline-induced Cardiac Toxicity; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Intervention Model Description: Randomization (1:1) will be stratified by LVEF on baseline CMR (as quantified by CMR core lab /CNIC), by research Centre and by patient's gender.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Conditioning (Active Comparator): Remote Ischemic Conditioning (RIC): Patients will undergo weekly RIC during the entire span of the chemotherapy period. Each RIC session will include four cycles of 5 min blood pressure cuff inflation followed by 5 min deflation
  Interventions: Device: RIPC
- simulated RIPC (Sham) (Sham Comparator): Control group (Sham): Patients will undergo weekly simulated RIC (sham) during the entire span of the chemotherapy period. Each sham session will include four cycles of 5 min blood pressure cuff inflation followed by 5 min deflation.
  Interventions: Device: Simulated RIPC (Sham)

INTERVENTIONS:
Device: RIPC — The procedure will be performed by using an electric auto-control device (modified blood pressure monitor for remote ischemic conditioning, Seagull Healthcare Aps, Denmark) for Remote Ischemic Conditioning in the arm. During the inflation period, the blood pressure cuff is inflated to 200 mmHg to stop blood flow in the arm.
  Arms: Remote Ischemic Conditioning
Device: Simulated RIPC (Sham) — The procedure will be performed by using an electric auto-control device (modified blood pressure monitor for remote ischemic conditioning, Seagull Healthcare Aps, Denmark) for Remote Ischemic Conditioning in the arm. During the inflation period, the blood pressure cuff is inflated to a low pressure not stopping blood flow in the arm.
  Arms: simulated RIPC (Sham)

SUMMARY:
Multinational, prospective, proof of concept phase II, double-blinded, sham-controlled, randomized clinical trial (RCT) to evaluate the efficacy and safety of Remote Ischaemic PreConditioning (RIPC) in Lymphoma patients receiving anthracyclines.

DETAILED DESCRIPTION:
Multinational, prospective, proof of concept phase II, double-blinded, sham-controlled, randomized clinical trial (RCT) to evaluate the efficacy and safety of Remote Ischaemic PreConditioning (RIPC) in lymphoma patients receiving anthracyclines. Patients scheduled to undergo ≥5 chemotherapy cycles will be eligible. Patients fulfilling all inclusion and no exclusion criteria will be enrolled and undergo baseline Cardiac Magnetic Baseline (CMR), and high sensitivity troponin (hsTn) and NT-proBNP blood test. Patients with confirmed LVEF >40% by CMR will be randomized 1:1 to RIPC vs simulated RIPC (Sham). After the third chemotherapy cycle, a second CMR+ hsTn/ NT-proBNP will be performed for the validation of the early marker of cardiotoxicity. A third hsTn/ NT-proBNP blood test will be performed in the last chemotherapy cycle. Nine weeks after finishing chemotherapy, a last CMR+ hsTn/ NT-proBNP will be performed. Patients will be followed-up for clinical events at 6, 12, 18, 30 and 42 months until the last patient undergoes the final CMR. When the last patient undergoes the third CMR, the follow-up will be closed. The median follow-up estimation for clinical endpoints is 36 months (range: 6 to 60 months).

ELIGIBILITY:
Inclusion Criteria:

≥18 years old NHL, HL or breast cancer diagnosis Scheduled to undergo chemotherapy including ≥ 240 mg/k2 cumulative dose of anthracyclines.

Pre-chemo LVEF >40% on screening echocardiography.

Presence of ≥1 of the following risk factors for developing cardiotoxicity:

Previous coronary artery disease (any of the following):

Previous coronary revascularisation (PCI or CABG) or Medical history of previous significant nonrevascularized coronary stenosis Previous Acute Coronary Syndrome / Acute Myocardial Infarction with a LVEF > 40 LVEF 41-54% Age ≥ 65 years old Previous diagnosis of arterial hypertension (with or without treatment) Chronic kidney disease (estimated glomerular filtration rate <60ml/min/1.73m2) Current or former smoker. Obesity (BMI≥30 kg/m2) LVH on screening echocardiography (LV thickness ≥12mm). High alcohol intake (≥21 alcoholic beverages per week) Sinus rhythm on screening ECG Previous diagnosis of diabetes (except those treated with sulfonylureas or those with neuropathy) Previous non-anthracycline-based chemotherapy Signed Informed Consent Form (ICF)

Exclusion Criteria:

* History of any of the following diseases:

  * Any cancer who received anthracyclines treatment before the index episode.
  * Previous clinical diagnosis of heart failure.
  * Permanent atrial fibrillation (AF).
  * Severe valvular or sub-valvular heart disease.
  * Severe peripheral arterial disease in the upper extremities or arteriovenous (AV) shunt in the arm selected for RIPC.
* Clinical diagnosis of diabetes neuropathy
* Contraindication for CMR:

  * Severe claustrophobia.
  * Any device which is known to threaten or pose hazard in all MR environments (http://www.mrisafety.com/).
  * Patients with implanted biomedical cardiac devices: pacemakers, ICDs or CRT.
* Severe thrombocytopenia (platelets <50,000/µL) on any blood test within the previous 3 months.
* Patients participating in other clinical trials.
* Impossibility to consent or undergo study follow-ups.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of anthracycline-induced cardiotoxicity events | 9 weeks after the last chemotherapy cycle (anticipated to be between 150 and 200 days from enrollment)
  Cardiotoxicity event is defined as one of the following:
  * Drop in LVEF between study CMRs of ≥10 absolute points regardless the absolute value of follow- up ejection fraction (EF).
  * Drop in LVEF between study CMRs of ≥5 to <10 absolute points with a follow-up EF value <50%
  UNITS: absolute number of patients in each arm qualifying for cardiotoxicity event (i.e. each patient will be qualified at the end of the study as YES/NO).

SECONDARY OUTCOMES:
Primary efficacy endpoint: (RIC vs Sham) Absolute change in LVEF | 9 weeks after the last chemotherapy cycle (anticipated to be between 150 and 200 days from enrollment)
  change in LVEF between baseline and any follow-up CMRs, whichever shows worse LVEF
  UNITS: LVEF is expressed as % LVEF= (LV end-diastolic volume - LV end-systolic volume) / LV end-systolic volume), %
Rate of tumor regression. | 9 weeks after the last chemotherapy cycle (anticipated to be between 150 and 200 days from enrollment)
  Response to chemotherapy
  UNITS: absolute number of patients in each arm qualifying as responder or no responder (i.e. each patient will be qualified at the end of the study as YES/NO).
Change in Quality of Life-Haematological Malignancy Patient-Reported Outcome Measure questionnaire | 9 weeks after the last chemotherapy cycle (anticipated to be between 150 and 200 days from enrollment)
  Haematological Malignancy Patient-Reported Outcome Measure (HM-PRO) questionnaire
  UNITS: absolute points in the questionnaire. minimum value 0 maximum value 84
  the higher the total score, the better (greater the effect on a patient's QoL)
Change in Quality of Life-Euro Quality of Life-5 dimensions questionnaire | 9 weeks after the last chemotherapy cycle (anticipated to be between 150 and 200 days from enrollment)
  Euro Quality of Life-5 dimensions (EuroQoL-5D) questionnaire:
  UNITS: absolute points in the questionnaire. minimum value 0 maximum value 100
  the higher the total score, the better (greater the effect on a patient's QoL)
Change in Quality of Life-Kansas City Cardiomyopathy Questionnaire | 9 weeks after the last chemotherapy cycle (anticipated to be between 150 and 200 days from enrollment)
  Kansas City Cardiomyopathy Questionnaire (KCCQ-12)
  UNITS: absolute points in the questionnaire. minimum value 0 maximum value 65
  the higher the total score, the better (greater the effect on a patient's QoL)
Rate of Heart Failure Hospitalization | 4-60 months
  Rate of Heart Failure Hospitalization
  UNITS: Absolute number of patients in each arm experiencing a heart failure hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Borja Ibañez, MD PhD FESC, Principal Investigator — CNIC
Locations (24):
- Aarhus University, Aarhus, Denmark
- France (2):
  - Hospital Jaques Monod, El Havre, Montivilliers
  - Henri Becquerel, Rouen
- University Hospital Duesseldorf UDUS, Düsseldorf, Germany
- Amsterdam UMC, Amsterdam, Netherlands
- Portugal (2):
  - Hospital da Luz Learning Health (GLSMED), Lisbon
  - IPO Lisboa, Lisbon
- Spain (17):
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares
  - Centro Medico Teknon, Barcelona
  - Instituto Catalán de Oncología, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Centro Nacional de Investigaciones Cardiovasculares (CNIC), Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario la Paz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Ruber Juan Bravo, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clinico Universitario de Valladolid, Valladolid

REFERENCES:
- See also: web page — http://resilience-h2020.com